CLINICAL TRIAL: NCT00723112
Title: The Role of Erythropoietin in Myelodysplastic Syndrome
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Josef T. Prchal, MD, University of Utah
Other Study IDs: 20716; DK007115-31
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; Erythropoiesis; Ineffective Hematopoiesis; Erythroid Progenitors; Dyserythropoiesis
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Affected Group: Adult subjects with the diagnosis of MDS based on the French-American-British classification system.
- Healthy Controls: Control subjects will be selected using frequency matching on gender and age by decade. That is for each MDS patient a healthy volunteer of the same gender and decade (50-59, 60-69, 70-79, etc) will be selected

SUMMARY:
The purpose of the study is to elucidate the causative molecular events responsible for the abnormal erythropoiesis in MDS.

DETAILED DESCRIPTION:
Myelodysplastic syndromes are a heterogeneous group of disorders characterized by clonal expansion of hematopoietic stem cells and ineffective hematopoiesis. Although all 3 cell lineages in myeloid hematopoiesis can be involved, the erythroid dysplasia and ineffective erythropoiesis of MDS are usually the most severe, and often precede the development of other bone marrow lineage defects.

In normal erythropoiesis, erythroid progenitors differentiate and proliferate in response to stimulation by erythropoietin (Epo). Epo binds to its receptor, EpoR, constitutively expressed at the surface of committed erythroid progenitors and induces homodimerization. This study is designed to evaluate the EpoR cDNA sequence and its level of expression in the clonal erythroid progenitors of MDS patients (in cells stratified for the same degree of erythroid maturation) to determine whether mutations in the EpoR may be responsible for an aberrant Epo signal transduction in MDS. As well as analyze intrinsic erythroid Epo expression to determine whether it differs between normal controls and patients with MDS and perform a microarray analysis of genes associated with Epo signal transduction to determine if MDS patients have abnormal expression of signal transduction proteins.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects greater than 18 years of age
* Diagnosis of MDS based on the French-American-British classification system (including secondary causes of MDS)

Exclusion Criteria:

* Subjects not meeting the criteria listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with myelodysplastic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2007-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the EpoR cDNA sequence and its level of expression in the clonal erythroid progenitors of MDS patients to determine whether mutations in the EpoR may be responsible for an aberrant Epo signal transduction in MDS. | After Samples are obtained

SECONDARY OUTCOMES:
Analyze intrinsic erythroid Epo expression to determine whether it differs between normal controls and patients with MDS. | After samples are obtained
Perform a microarray analysis of genes associated with Epo signal transduction to determine if MDS patients have abnormal expression of signal transduction proteins. | After samples are obtained
Determine how often and what percent clonality occurs in MDS patients and try to predict who has early MDS by clonality testing. | After samples from female patients have been obtained

CONTACTS AND LOCATIONS:
Overall Officials: Josef T Prchal, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - VA Salt Lake City Health Care System, Salt Lake City, Utah

REFERENCES:
- [Background] Aul C, Arning M, Runde V, Schneider W. Serum erythropoietin concentrations in patients with myelodysplastic syndromes. Leuk Res. 1991;15(7):571-5. doi: 10.1016/0145-2126(91)90025-o. PMID 1861540
- [Background] Stasi R, Brunetti M, Terzoli E, Abruzzese E, Amadori S. Once-weekly dosing of recombinant human erythropoietin alpha in patients with myelodysplastic syndromes unresponsive to conventional dosing. Ann Oncol. 2004 Nov;15(11):1684-90. doi: 10.1093/annonc/mdh428. PMID 15520072
- [Background] Casadevall N, Durieux P, Dubois S, Hemery F, Lepage E, Quarre MC, Damaj G, Giraudier S, Guerci A, Laurent G, Dombret H, Chomienne C, Ribrag V, Stamatoullas A, Marie JP, Vekhoff A, Maloisel F, Navarro R, Dreyfus F, Fenaux P. Health, economic, and quality-of-life effects of erythropoietin and granulocyte colony-stimulating factor for the treatment of myelodysplastic syndromes: a randomized, controlled trial. Blood. 2004 Jul 15;104(2):321-7. doi: 10.1182/blood-2003-07-2252. Epub 2004 Mar 30. PMID 15054036
- [Background] Solignac M; European Hematology Association. [Epoetin beta, new strategies to optimise the management of anaemia in cancer patients]. Presse Med. 2003 Sep 13;32(29):1385-8. No abstract available. French. PMID 14534506
- [Background] Fontenay-Roupie M, Bouscary D, Guesnu M, Picard F, Melle J, Lacombe C, Gisselbrecht S, Mayeux P, Dreyfus F. Ineffective erythropoiesis in myelodysplastic syndromes: correlation with Fas expression but not with lack of erythropoietin receptor signal transduction. Br J Haematol. 1999 Aug;106(2):464-73. doi: 10.1046/j.1365-2141.1999.01539.x. PMID 10460607
- [Background] Takeshita A, Shinjo K, Naito K, Ohnishi K, Higuchi M, Ohno R. Erythropoietin receptor in myelodysplastic syndrome and leukemia. Leuk Lymphoma. 2002 Feb;43(2):261-4. doi: 10.1080/10428190290006026. PMID 11999556
- [Background] Shinjo K, Takeshita A, Higuchi M, Ohnishi K, Ohno R. Erythropoietin receptor expression on human bone marrow erythroid precursor cells by a newly-devised quantitative flow-cytometric assay. Br J Haematol. 1997 Mar;96(3):551-8. doi: 10.1046/j.1365-2141.1997.d01-2071.x. PMID 9054663
- [Background] McMullin MF, Percy MJ. Erythropoietin receptor and hematological disease. Am J Hematol. 1999 Jan;60(1):55-60. doi: 10.1002/(sici)1096-8652(199901)60:13.0.co;2-v. PMID 9883806
- [Background] Kralovics R, Sokol L, Broxson EH Jr, Prchal JT. The erythropoietin receptor gene is not linked with the polycythemia phenotype in a family with autosomal dominant primary polycythemia. Proc Assoc Am Physicians. 1997 Nov;109(6):580-5. PMID 9394420
- [Background] Kralovics R, Indrak K, Stopka T, Berman BW, Prchal JF, Prchal JT. Two new EPO receptor mutations: truncated EPO receptors are most frequently associated with primary familial and congenital polycythemias. Blood. 1997 Sep 1;90(5):2057-61. PMID 9292543
- [Background] Stopka T, Zivny JH, Stopkova P, Prchal JF, Prchal JT. Human hematopoietic progenitors express erythropoietin. Blood. 1998 May 15;91(10):3766-72. PMID 9573013
- [Background] Sato TN. A new role of lipid receptors in vascular and cardiac morphogenesis. J Clin Invest. 2000 Oct;106(8):939-40. doi: 10.1172/JCI11304. No abstract available. PMID 11032853